CLINICAL TRIAL: NCT03297463
Title: A Phase 1b/2 Study of Hypofractionated Radiation and Combination Immunotherapy for Relapsed/Refractory Metastatic Melanoma
Brief Title: Radiation Therapy With Combination Immunotherapy for Relapsed/Refractory Metastatic Melanoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Replaced by another study.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS172
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Melanoma; Pulmonary Metastases; Hepatic Metastases; Brain Metastases
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Interleukin-2; Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase Ib (Dose Escalation) (Experimental)
  Interventions: Drug: Interleukin-2 & Ipilimumab (P-Ib)
- Phase II (Dose Expansion) (Experimental)
  Interventions: Drug: Interleukin-2 & Ipilimumab (P-II)

INTERVENTIONS:
Drug: Interleukin-2 & Ipilimumab (P-Ib) — Phase Ib:
  - Ipilimumab will be administered in a 3 + 3 dose escalation design.
  * The starting dose will be 0.3 mg/kg administered within 7 days of day 1 cycle 2 ALdesleukin (IL-2).
  * If dose limiting autoimmune toxicities (DLTs) are not observed, the next cohort will receive 1.5 mg/kg.
  * The final cohort will receive 3 mg/kg, in the event that cohort 2 does not exhibit DLTs.
  * In the event of excessive toxicity in cohort 1, then a -1 dose level of 0.1 mg/kg may be evaluated in subsequent cohorts. Cohort sizes will increase to 6 patients if 1 of 3 patients in a cohort experience a DLT.
  * Once the maximum tolerated dose/recommended phase 2 dose (MTD/RP2D) is declared, no staggering of enrollment is required for accrual.
  Other Names: IL-2; Yervoy
  Arms: Phase Ib (Dose Escalation)
Drug: Interleukin-2 & Ipilimumab (P-II) — Phase II:
  - Interleukin-2 & Ipilimumab will be administered at the maximum tolerated dose/recommended phase 2 dose (MTD/RP2D).
  Other Names: IL-2; Yervoy
  Arms: Phase II (Dose Expansion)

SUMMARY:
This is a Phase 1b/2 study designed to evaluate combination of the human T-cell cytokine Interleukin-2 (IL-2) and a checkpoint inhibitor Ipilimumab immediately following a course of hypofractionated palliative radiation therapy in the management of unresectable, relapsed/refractory metastatic melanoma.

DETAILED DESCRIPTION:
The sequential administration of Interleukin-2 (IL-2) following radiation therapy offers a rational immunologic priming strategy to expand antigen primed T cells under the growth promoting effects of Interleukin-2 therapy.

This clinical trial is designed to evaluate the combination of the T cell cytokine Interleukin-2 and the checkpoint inhibitor Ipilimumab in sequential combination following a course of hypofractionated palliative radiation therapy. The addition of single dose Ipilimumab offers rational timing of CTLA-4 checkpoint blockade to decrease activity of regulatory and suppressor T cell subsets following IL-2 based immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven unresectable, metastatic melanoma refractory to standard immunotherapy drugs or regimens, including prior treatment with Aldesleukin (IL-2), GM-CSF, Ipilimumab, Nivolumab, Pembrolizumab, and/or Imlygic (T-VEC).
* Prior clinical trial participation or treatment with molecularly targeted agents (i.e. Vemurafenib/Cobimetinib, Dabrafenib/Trametinib) or chemotherapy (i.e. Temozolomide, Dacarbazine, Platinum, or Taxanes) is permitted.
* Must have a minimum of 3 radiographically distinct (>1.5 cm) lesions measurable by RECIST 1.1 at time of study enrollment (>5 preferred).

  * A maximum of 2 metastases per treated organ may be targeted for HD-XRT, but must be separated by more than 5 cm of normal tissue
  * At least 2 non-irradiated lesions are required for systemic response assessments
* Pulmonary metastases: Pulmonary metastasis permissible. Appropriate candidates with lung lesions may be considered for ablative hypofractionation using SBRT.
* Hepatic metastases: Hepatic metastasis permissible. Appropriate candidates with metastasis to liver may be considered for ablative hypofractionation using SBRT.
* Brain metastases: Brain metastases may be treated using Gamma Knife Radiosurgery (GKR) or whole brain radiation therapy (WBRT) per the treating radiation oncologist. Total radiation dose and number of fractions will be determined by the treating radiation oncologist based on anatomic and dosing constraints. MRI of the vertebral column is required for all patients with suspected epidural tumor extension.
* Must have sufficient archival tissue block material (1.5 x 1.5 x 1.5 cm) and/or newly obtained core or excisional biopsy of tumor tissue; minimum of 2 cores.
* ECOG performance status 0 or 1 (appendix 2)
* Age 18 to 85 years of age; > 85 years of age must be approved by Principal Investigator.
* Adequate organ function within 14 days of registration (30 days for pulmonary and cardiac assessments) defined as:

  * Hematologic: Leukocytes ≥ 3,000/mcL, ANC ≥ 1,000/mcL, Hemoglobin ≥ 9.0 g/dL, Platelets ≥ 120,000/mcL
  * Renal: Serum creatinine ≤ 1.8 mg/dL; for patients with a creatinine > 1.5 mg/dL or a history of renal dysfunction, an estimated glomerular filtration rate ≥ 35 mL/min/1.73 m2 is required
  * Hepatic: AST, ALT, and alkaline phosphatase ≤ 10 x upper limit of normal and total bilirubin ≤ 2.0 mg/dL Pulmonary: oxygen saturation ≥90% on room air; corrected DLCO and FEV1, ≥ 50% predicted
  * Cardiac: Absence of clinical decompensated congestive heart failure or uncontrolled arrhythmia; left ventricular ejection fraction (echocardiogram within 6 months permitted) ≥ 40%. QTc must be < 450 ms in males and < 470 ms in females.
* Time from last anti-tumor treatment to first radiation treatment at least 1 week.
* Recovery from previous cancer treatment (≤ Grade 1 by CTCAE 4.0 criteria) prior to first radiation treatment
* Women of childbearing potential and males with partners of childbearing potential must agree to the use of barrier methods of contraception, hormonal contraceptives, or to abstain from heterosexual activity for the duration of study participation.
* Ability to understand and provide voluntary written informed consent

Exclusion Criteria:

* Pregnant or breast feeding. The agents used in this study have the potential to harm a fetus. Radiation is a known teratogen. There is insufficient information regarding potential for fetal harm during immunotherapy at this time. Biological females of childbearing potential must have a negative serum pregnancy test within 14 days of registration.
* Diagnosis of immunodeficiency
* Concurrent use of high dose steroids; chronic steroid use of < 2 mg dexamethasone or equivalent per day is permissible
* Concurrent malignancy requiring active treatment, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ
* Prior organ allograft or allogeneic transplantation
* Autoimmune disease
* Uncontrolled intercurrent or psychiatric illness or social situation that would limit compliance with study requirements
* Live vaccines within 30 days prior to the first dose of IL-2 and while participating in the trial. Examples of live vaccines include, but are not limited to, measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed. However, intranasal influenza vaccines (eg, Flu - Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose (MTD) | Cycle 2 Day 1
  Incidence of Adverse Events
Phase 1: Maximum Tolerated Dose (MTD) | Cycle 2 Day 15
  Incidence of Adverse Events
Phase 1: Maximum Tolerated Dose (MTD) | 30 days after last IL-2
  Incidence of Adverse Events
Phase 2: Objective Response Rate (ORR) | Day 35
  Disease re-assessment includes physical examination, as well as radiographic response assessment (RECIST v1.1) of non-irradiated target lesions using CT (or PET/CT) and/or at MRI.
Phase 2: Objective Response Rate (ORR) | 30 days after last IL-2
  Disease re-assessment includes physical examination, as well as radiographic response assessment (RECIST v1.1) of non-irradiated target lesions using CT (or PET/CT) and/or at MRI.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Every 3 Months until 2 Years from 1st IL-2 Dose
  Incidence of PFS
Overall survival (OS) | Every 3 Months until 2 Years from 1st IL-2 Dose
  Incidence of OS

CONTACTS AND LOCATIONS:
Overall Officials: Domingo-Musibay Evidio, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center - University of Minnesota, Minneapolis, Minnesota, United States